CLINICAL TRIAL: NCT00721760
Title: A Multinational, Multicenter, Randomized, Double-Blind Study Comparing the Efficacy and Safety of AVE5026 With Enoxaparin for the Prevention of Venous Thromboembolism in Patients Undergoing Hip Fracture Surgery
Brief Title: Evaluation of AVE5026 as Compared to Enoxaparin for the Prevention of Thromboembolism in Patients Undergoing Hip Fracture Surgery
Acronym: SAVE-HIP2
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: EFC10343; 2007-007945-11 (EudraCT Number)
Record Dates: First submitted 2008-07-22; First posted 2008-07-24 (Estimated); Last update posted 2013-01-23 (Estimated); Status verified 2013-01

CONDITIONS: Venous Thromboembolism
Keywords: Hip fractures; Heparin Low-Molecular-Weight; Randomized Controlled Trial
MeSH Terms: conditions — Venous Thromboembolism; Hip Fractures | interventions — enoxaparin sodium; Enoxaparin; AVE 5026

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Semuloparin (Experimental): Semuloparin sodium 20 mg (10 mg if Severe Renal Impairment [SRI]) once daily for 7-10 days with an initial dose given 8 hours after surgery
  Placebo for Enoxaparin sodium prior to surgery according to local standard for Enoxaparin and 12 hours after surgery to maintain the blind
  Interventions: Drug: Semuloparin sodium; Drug: Placebo
- Enoxaparin (Active Comparator): Enoxaparin sodium 40 mg (20 mg if Severe Renal Impairment [SRI]) once daily for 7-10 days with an initial dose given prior to or 12 hours after surgery according to local standard for Enoxaparin sodium
  Placebo for Semuloparin sodium 8 hours after surgery to maintain the blind
  Interventions: Drug: Enoxaparin sodium; Drug: Placebo

INTERVENTIONS:
Drug: Enoxaparin sodium — 0.4 mL (0.2 mL if SRI) solution in ready-to-use 0.5 ml pre-filled syringe
  Subcutaneous injection
  Other Names: Lovenox®
  Arms: Enoxaparin
Drug: Semuloparin sodium — 0.4 mL (0.2 mL if SRI) solution in ready-to-use 0.5 ml pre-filled syringe
  Subcutaneous injection
  Other Names: AVE5026
  Arms: Semuloparin
Drug: Placebo — 0.4 mL (0.2 mL if SRI) solution in ready-to-use 0.5 ml prefilled syringe strictly identical in appearance but without active component
  Subcutaneous injection

SUMMARY:
The primary objective was to compare the efficacy of once daily [q.d] subcutaneous [s.c.] injections of Semuloparin sodium (AVE5026) with q.d. s.c. injections of Enoxaparin for the prevention of Venous Thromboembolic Events [VTE] in patients undergoing hip fracture surgery.

The secondary objectives were to evaluate the safety of AVE5026 in patients undergoing hip fracture surgery, and to document AVE5026 exposure in this population.

DETAILED DESCRIPTION:
Randomization had to take place just prior to the first study drug injection (randomization ratio 1:1).

The total duration of observation per participant was 35-42 days from surgery broken down as follows:

* 7 to 10-day double-blind treatment period;
* 28 to 35-day follow-up period.

Mandatory bilateral venography of the lower limbs had to be performed between 7 to 11 days after surgery.

ELIGIBILITY:
Inclusion Criteria:

* Standard surgery for fracture of the upper third of the femur including femoral head and neck.

Exclusion Criteria:

* Estimated time of injury/fracture > 24 hours before admission to hospital;
* Any major orthopedic surgery in the 3 months prior to study start;
* Multiple trauma affecting more than one organ system;
* Deep vein thrombosis or pulmonary embolism within the last 12 months or known post-phlebitic syndrome;
* High risk of bleeding;
* Known allergy to heparin, or enoxaparin, or pork products;
* End stage renal disease or patient on dialysis;

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1003 (Actual)
Dates: Start 2008-07; Primary Completion 2009-10 (Actual); Study Completion 2009-10 (Actual)

PRIMARY OUTCOMES:
Percentage of Participants Who Experienced Venous Thromboembolism Event [VTE] or All-cause Death | From randomization up to 10 days after surgery or the day of mandatory venography, whichever came first
  VTE included any Deep Vein Thrombosis [DVT] (proximal or distal, symptomatic or not) and non-fatal Pulmonary Embolism [PE] as confirmed by a Central Independent Adjudication Committee [CIAC] after review of mandatory bilateral venograms and diagnostic tests for VTE.
  All-cause deaths included fatal PE and deaths for other reason than PE.

SECONDARY OUTCOMES:
Percentage of Participants Who Experienced "Major" VTE or All-cause Death | From randomization up to 10 days after surgery or the day of mandatory venography, whichever came first
  "major" VTE included any proximal DVT, symptomatic distal DVT and non-fatal PE as confirmed by the CIAC.
Percentage of Participants Who Experienced Clinically Relevant Bleedings | From first study drug injection up to 3 days after last study drug injection
  Bleedings were centrally and blindly reviewed by the CIAC and classified as:
  * "major" (fatal, in a critical area/organ, causing a post-operative drop in hemoglobin ≥2 g/dL or requiring post-operative transfusion ≥2 units of blood, leading to an invasive diagnostic or therapeutic intervention, or associated with circulatory decompensation);
  * "clinically relevant non-major" (skin hematoma or epistaxis requiring surgical/medical intervention/treatment, macroscopic hematuria, or overt bleeding requiring specific attention by healthcare professional);
  * "Non-clinically relevant bleeding".
Percentage of Participants Who Required the Initiation of Curative Anticoagulant or Thrombolytic Treatment After VTE Assessment | From randomization up to 10 days after surgery or the day of mandatory venography, whichever came first
  Initiation of curative anticoagulant or thrombolytic treatment after VTE assessment was defined from investigator's answer to the question "was the subject treated for VTE?" asked after the diagnostic tests for suspected VTE and after the mandatory venography.

OTHER OUTCOMES:
Overview of deaths | From first study drug injection up to 3 days after last study drug injection
  All deaths were centrally and blindly reviewed by the CIAC and classified as fatal PE, fatal bleeding, cardiovascular death or other based on relevant documentation (e.g. autopsy report).
Platelets Count: Percentage of Participants With Potentially Clinically Significant Abnormalities [PCSA] | From first study drug injection up to 3 days after last study drug injection
  PCSA are abnormal values considered medically important by the Sponsor according to predefined criteria based on literature review.
  Threshold for platelet counts was defined as <100 Giga/L.
Liver Function: Percentage of Participants With Potentially Clinically Significant Abnormalities [PCSA] | From first study drug injection up to 3 days after last study drug injection
  Thresholds were defined as follows:
  * Alanine Aminotransferase [ALAT] >3 Upper Normal Limit [ULN];
  * Total Bilirubin [TB] >2 ULN;
  * ALAT >3 ULN and TB >2 ULN;
  Cases with ALAT >3 ULN and TB >2 ULN (not necessarily concomitant) were evaluated by a blinded independent adjudicator to determine if they met Hy's law criteria.

CONTACTS AND LOCATIONS:
Overall Officials: William D. Fisher, MD, Principal Investigator — Department of Orthopaedic Surgery, McGill University Health Centre, 1650 Cedar Avenue, Montreal, Quebec, H3G 1A4, Canada; Alexander G. Turpie, Study Chair — McMaster University
Locations (25):
- Sanofi-Aventis Administrative Office, Bridgewater, New Jersey, United States
- Sanofi-Aventis Administrative Office, Buenos Aires, Argentina
- Sanofi-Aventis Administrative Office, Minsk, Belarus
- Sanofi-Aventis Administrative Office, Sofia, Bulgaria
- Sanofi-Aventis Administrative Office, Laval, Canada
- Sanofi-Aventis Administrative Office, Santiago, Chile
- Sanofi-Aventis Administrative Office, Shangaï, China
- Sanofi-Aventis Administrative Office, Bogotá, Colombia
- Sanofi-Aventis Administrative Office, Prague, Czechia
- Sanofi-Aventis Administrative Office, Hørsholm, Denmark
- Sanofi-Aventis Administrative Office, Helsinki, Finland
- Sanofi-Aventis Administrative Office, Athens, Greece
- Sanofi-Aventis Administrative Office, Mumbai, India
- Sanofi-Aventis Administrative Office, Milan, Italy
- Sanofi-Aventis Administrative Office, México, Mexico
- Sanofi-Aventis Administrative Office, Lima, Peru
- Sanofi-Aventis Administrative Office, Warsaw, Poland
- Sanofi-Aventis Administrative Office, Porto Salvo, Portugal
- Sanofi-Aventis Administrative Office, Bucharest, Romania
- Sanofi-Aventis Administrative Office, Moscow, Russia
- Sanofi-Aventis Administrative Office, Midrand, South Africa
- Sanofi-Aventis Administrative Office, Barcelona, Spain
- Sanofi-Aventis Administrative Office, Bromma, Sweden
- Sanofi-Aventis Administrative Office, Istanbul, Turkey (Türkiye)
- Sanofi-Aventis Administrative Office, Kiev, Ukraine

REFERENCES:
- [Result] Lassen MR, Fisher W, Mouret P, Agnelli G, George D, Kakkar A, Mismetti P, Turpie AG; SAVE Investigators. Semuloparin for prevention of venous thromboembolism after major orthopedic surgery: results from three randomized clinical trials, SAVE-HIP1, SAVE-HIP2 and SAVE-KNEE. J Thromb Haemost. 2012 May;10(5):822-32. doi: 10.1111/j.1538-7836.2012.04701.x. PMID 22429800